CLINICAL TRIAL: NCT04733027
Title: Dose Escalation, First-in-human Clinical Trial to Evaluate the Safety, Pharmacokinetics and Preliminary Antitumor Activity of PEP-010, Administered as Single Agent and in Combination With Paclitaxel or With Gemcitabine in Patients With Metastatic Solid Cancer
Brief Title: First-in-human Phase I to Evaluate PEP-010 as Single Agent and in Combination With Paclitaxel or With Gemcitabine (CleverPeptide)
Acronym: Clever Peptide
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IC 2018-06
Record Dates: First submitted 2021-01-22; First posted 2021-02-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Solid Tumor Cancer

STUDY DESIGN:
Intervention Model Description: Part 1 dose escalation Part 2 expansion cohort and short dose escalation cohort Randomization in the escalation dose cohort once MTD defined
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 2 cohort 1 : PEP010 in combination with paclitaxel (Experimental): Fort part 2 the Cohort 1 will include patients with PDAC treated with the combination of PEP-010 at the dose of 2.5 mg/kg and weekly paclitaxel 80 mg/m².
  Interventions: Combination Product: Dose escalation, first-in-human phase I clinical trial with an Expansion phase
- Part 2 cohort 2 : PEP010 in combination with gemcitabine (Experimental): In arm B, the dose escalation phase will begin with DL4 (1.2 mg/kg) and will follow a 3+3 design For part 2 Cohort 2 will include patients with PDAC or OC treated with the combination of PEP-010 in ascending doses, and gemcitabine at 1000 mg/m2.
  Four doses of PEP-010 will be tested: 1.2 mg/kg, 2.5 mg/kg, 5 mg/kg and 10 mg/kg, according to a 3+3 dose escalation design.
  Once a MTD is achieved, and in light of safety, PK, and PD data, two dosing schedules will be further explored based on TSC recommendations. Each dosing schedule will be evaluated in a separate cohort to generate more data and inform on the choice of the RP2D, as per the recommendations of the FDA (Project Optimus). Patients will be randomized simultaneously in the two dose cohorts, each would include approximately 6 - 10 patients.
  Interventions: Combination Product: Dose escalation, first-in-human phase I clinical trial with an Expansion phase

INTERVENTIONS:
Combination Product: Dose escalation, first-in-human phase I clinical trial with an Expansion phase — PEP-010 will be administered on days 1, 2 and 3 every week, as a 3-hour intravenous infusion. Treatment will be administered until disease progression, unacceptable toxicity, death or withdrawal of consent, whichever occurs first. Each cycle will be of 21 days duration.

SUMMARY:
This is an open-label, non-controlled, multicenter, dose escalation, first-in-human phase I clinical trial with an expansion phase designed to assess the safety, tolerability, PK and PD parameters, and preliminary antitumor activity of intravenous dosing of PEP-010 as single agent and in combination with paclitaxel or with gemcitabine

PEP-010 will be administered, in a Part 1, as single agent in patients with solid cancers who are not amenable to standard treatment, or in combination in patients who are eligible for the paclitaxel therapy, and in a Part 2 only in combination in:

Cohort 1 (expansion cohort, phase 1b): metastatic pancreatic ductal carcinoma (PDAC) who received at least one previous systemic chemotherapy and eligible for paclitaxel therapy.

Cohort 2 (dose escalation cohort, phase 1a): metastatic pancreatic ductal carcinoma or advanced/metastatic ovarian cancer (OC) eligible for gemcitabine-based therapy

DETAILED DESCRIPTION:
Part 1 : PEP-010 was administered on days 1, 2 and 3 every week. Treatment was administered until disease progression, unacceptable toxicity, death or withdrawal of consent, whichever occured first. Each cycle was of 21 days duration.

The initial starting dose of PEP-010, DL1 was selected based on pre-clinical data at 0.15 mg/kg. The other doses per injection from DL2 to DL7 are 0.3, 0.6; 1.2; 2.5; 5; 10 and 15 mg/kg.

For patients in Arm B, PEP-010 was combined with Paclitaxel, at a dose of 80 mg/m², weekly until disease progression or unacceptable toxicity. Paclitaxel will be administered according to local guidelines.

Main objective for Dose escalation cohorts was to determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of PEP-010 when administered as single agent (MTD1/RP2D1), and in combination with paclitaxel (MTD2/RP2D2) by recording the dose-limiting toxicities (DLTs).

Secondary objectives were

* To evaluate the safety and tolerability of PEP-010 when administered as single agent, and in combination with paclitaxel.
* To assess the pharmacokinetics (PK) of PEP-010 as single agent, and in combination with paclitaxel in Dose escalation cohorts.
* To assess the pharmacodynamic (PD) effects of PEP-010 as single agent, and in combination with paclitaxel.
* To evaluate the preliminary antitumor activity of PEP-010 alone and in combination with paclitaxel, using Objective Response Rate (ORR), Progression-Free Survival (PFS) according to RECIST1.1, duration of response, and Overall Survival (OS).
* To assess the immunogenicity of PEP-010 as single agent, and in combination with paclitaxel in Dose escalation cohorts.

Part 2 :

In Part 2 - Cohort 1, PDAC patients will receive PEP-010 at dose 2.5 mg/kg in combination with paclitaxel administered at a dose of 80 mg/m² weekly.

In Part 2 - Cohort 2, PDAC and OC patients will receive PEP-010 at doses 1.2 to 10 mg/kg (short dose escamation) in combination with gemcitabine administered at a dose of 1000 mg/m² weekly during 3 weeks followed by a week without infusion.

Main objectives for Part 2 (Cohort 1)

• To determine the efficacy of PEP-010 in combination with paclitaxel in patients with pancreatic ductal adenocarcinoma by assessment of the objective response rate.

Part 2 (Cohort 2)

* To determine the MTD of PEP-010 when administered in combination with gemcitabine.
* To determine the RP2D of PEP-010 when administered in combination with gemcitabine.

Secondary objectives for Part 2 (Cohorts 1 and 2 )

* To evaluate the safety and tolerability of PEP-010 when administered in combination with paclitaxel or with gemcitabine.
* To complete the pharmacokinetics (PK) of PEP-010 in combination with paclitaxel.
* To assess the pharmacokinetics (PK) of PEP-010 in combination with gemcitabine.
* To assess the pharmacokinetics (PK) of paclitaxel, when administered in combination with PEP-010.
* To assess the pharmacokinetics (PK) of gemcitabine, when administered in combination with PEP-010.
* To characterize the PD effects of PEP-010 in combination with paclitaxel or with gemcitabine.
* To evaluate the preliminary antitumor activity of PEP-010 in combination with paclitaxel at the RP2D in term of PFS, duration of response and OS (Cohort 1).
* To evaluate the preliminary antitumor activity of PEP-010 in combination with gemcitabine using the ORR, PFS, duration of response and OS (Cohort 2).
* To assess the immunogenicity of PEP-010 in combination with paclitaxel or gemcitabine

ELIGIBILITY:
Inclusion criteria:

Part 1 Arms A and B:

1. Arm A: Patients must have histologically confirmed diagnosis of recurrent and/or metastatic solid tumors, who are not amenable to standard therapy, with exceptions as defined in the non-inclusion criteria,
2. Arm B: Patients must have histologically confirmed diagnosis of recurrent and/or metastatic solid tumors. Patients must be eligible for a treatment with paclitaxel as single agent. Patients who are eligible for standard of care paclitaxel-based combination therapy should not be included in the trial unless they have been previously exposed to that specific combination therapy. Specifically :

   * Patients with ovarian cancer must have received prior therapy with paclitaxel as part of standard of care in combination with carboplatin.
   * Patients with triple negative breast cancer are eligible for the trial since paclitaxel as single agent is standard of care in this disease.
3. Age ≥ 18 years,
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1,
5. Patients must have measurable disease (as per RECIST version 1.1),
6. Patient ability to comply with the collection of tumor biopsies, and tumors must be accessible for biopsy,
7. Adequate bone marrow function as defined by: Absolute Neutrophil Count (ANC) of ≥ 1.5 x 109/L, platelet count of ≥ 100 x 109/L, and hemoglobin of ≥ 9 g/dL),
8. Adequate liver function, as determined by a serum total bilirubin ≤ 1.5 Upper Limit of Normal (ULN), AST and ALT ≤ 3 x ULN (≤ 5 x ULN if liver metastases),
9. Adequate renal function, as determined by a serum creatinine ≤ 1.5 x ULN,
10. Provision of signed written informed consent,
11. Patient ability to comply with protocol requirements,
12. If the patient is female:

    * Patient must be postmenopausal, surgically sterile, or they must agree to use a physical barrier method of contraception in addition to either an intrauterine device or hormonal contraception until at least 6 months after termination of study drug or must refrain from heterosexual activity during this same period.
    * Patients of childbearing potential must have a negative pregnancy test within the seven days prior to the first study drug administration.

    If the patient is male:

    - Patient must abstain from heterosexual activity or must agree to use an acceptable method of contraception (e.g., condom) during the study for at least 6 months after termination of study drug.
13. Patients covered by a health insurance system;

Part 2 Cohort 1 Pancreatic Ductal adenocarcinoma (PDAC)

1. Age ≥ 18 years,
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1,
3. Patients must have measurable disease (as per RECIST version 1.1),
4. Patient ability to comply with the collection of tumor biopsies, and tumors must be accessible for biopsy,
5. Adequate bone marrow function as defined by: Absolute Neutrophil Count (ANC) of ≥ 1.5 x 109/L, platelet count of ≥ 100 x 109/L, and hemoglobin of ≥ 9 g/dL),
6. Adequate liver function, as determined by a serum total bilirubin ≤ 1.5 Upper Limit of Normal (ULN), AST and ALT ≤ 3 x ULN (≤ 5 x ULN if liver metastases),
7. Adequate renal function, as determined by a serum creatinine ≤ 1.5 x ULN,
8. Provision of signed written informed consent,
9. Patient ability to comply with protocol requirements,
10. If the patient is female:

    * Patient must be postmenopausal, surgically sterile, or they must agree to use a physical barrier method of contraception in addition to either an intrauterine device or hormonal contraception until at least 6 months after termination of study drug or must refrain from heterosexual activity during this same period.
    * Patients of childbearing potential must have a negative pregnancy test within the seven days prior to the first study drug administration.

    If the patient is male:

    - Patient must abstain from heterosexual activity or must agree to use an acceptable method of contraception (e.g., condom) during the study for at least 6 months after termination of study drug.
11. Patients covered by a health insurance system
12. Histologically confirmed metastatic pancreatic ductal adenocarcinoma (mixed histology is acceptable as long adenocarcinoma is the dominant histological subtype)
13. Patient should have received at least one previous line of systemic treatment in metastatic setting
14. No previous disease progression under taxane therapy or 12-month free interval since last taxane therapy.

Part 2 Cohort 2 Pancreatic Ductal adenocarcinoma (PDAC) or Ovarian Cancer (OC)

1. Age ≥ 18 years,
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1,
3. Patients must have measurable disease (as per RECIST version 1.1),
4. Patient ability to comply with the collection of tumor biopsies, and tumors must be accessible for biopsy,
5. Adequate bone marrow function as defined by: Absolute Neutrophil Count (ANC) of ≥ 1.5 x 109/L, platelet count of ≥ 100 x 109/L, and hemoglobin of ≥ 9 g/dL),
6. Adequate liver function, as determined by a serum total bilirubin ≤ 1.5 Upper Limit of Normal (ULN), AST and ALT ≤ 3 x ULN (≤ 5 x ULN if liver metastases),
7. Adequate renal function, as determined by a serum creatinine ≤ 1.5 x ULN,
8. Provision of signed written informed consent,
9. Patient ability to comply with protocol requirements,
10. If the patient is female:

    * Patient must be postmenopausal, surgically sterile, or they must agree to use a physical barrier method of contraception in addition to either an intrauterine device or hormonal contraception until at least 6 months after termination of study drug or must refrain from heterosexual activity during this same period.
    * Patients of childbearing potential must have a negative pregnancy test within the seven days prior to the first study drug administration.

    If the patient is male:

    - Patient must abstain from heterosexual activity or must agree to use an acceptable method of contraception (e.g., condom) during the study for at least 6 months after termination of study drug.
11. Patients covered by a health insurance system
12. Patient must be eligible but not previously treatment with gemcitabine.

    Specific Pancreatic Ductal adenocarcinoma (PDAC)
13. Histologically confirmed metastatic pancreatic ductal adenocarcinoma (mixed histology is acceptable as long adenocarcinoma is the dominant histological subtype)

    Specific ovarian cancer (OC)
14. Patient has been diagnosed with recurrent epithelial ovarian, peritoneal, or fallopian tube carcinoma.
15. Subjects had disease recurrence or progression during prior chemotherapy with platinum-based regimens or within 6 months after the last dose of chemotherapy with platinum-based regimens (for at least 4 cycles of treatment)
16. Patient should have received at least one previous line of treatment in platinum-resistant setting.

Non-inclusion criteria: Part 1 Arms A and B, Part 2 Cohorts 1 and 2

1. Arm B and Cohort 1: Allergy or hypersensitivity to paclitaxel or components of the paclitaxel formulation,
2. Cohort 2: Allergy or hypersensitivity to gemcitabine or components of the gemcitabine formulation,
3. Allergy or hypersensitivity to PEP-010 formulation (Trehalose, Tween 20),
4. Patients with known or suspected Central Nervous System (CNS) metastases including leptomeningeal metastasis (except patients with radiographically stable, asymptomatic previously irradiated lesion provided patient is ≥ 3 weeks beyond completing cranial irradiation),
5. Evidence of significant, uncontrolled concomitant diseases, which could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina), or pulmonary disease (including obstructive pulmonary disease and history of symptomatic bronchospasm),
6. Concomitant cancer in the past 3 years except prostate cancer controlled by hormone therapy, cutaneous cancers (except melanoma) and in situ carcinoma,
7. Prior chemotherapy, radiotherapy (other than short cycle of palliative radiotherapy), immunotherapy within 21 days of first receipt of study drug,
8. Prior investigational agent within 28 days of first PEP-010 administration,
9. Hormone therapy within 14 days of first receipt of study drug, with exception of Gonadotropin-Releasing Hormone (GnRH) or Luteinizing-Hormone-Releasing Hormone (LHRH) agonists used for advanced prostate cancer, if indicated,
10. Prior relevant toxicities from chemotherapy or radiotherapy which have not regressed to grade ≤1 severity except alopecia (NCI-CTCAE version 5.0),
11. Patients with acute infection.
12. Any other uncontrolled diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding or any other medical condition that, in the opinion of the investigator, contraindicates the use of an investigational drug, or will impose excessive risk to the patient,
13. Patients with known HIV, HBV and HCV infections,
14. Patients with known active Sars Cov 2 infection
15. Pregnant or lactating women,
16. Patients with altered mental status or psychiatric disorder that, in the opinion of the investigator, would preclude a valid patient informed consent,
17. Person deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
For Part 1 (Dose escalation) and Part 2 (Cohort 2), the primary endpoints are the rate of occurrence of DLT within cycle 1 (21 days) after initiation of the study treatment for both parts. | 21 days after study treatment initiation
  The DLT is defined as any clinically significant non-hematological toxicity ≥ grade 3 and any hematological toxicity ≥ grade 4 of treatment-related adverse event
Part 2 Cohort 1: The primary endpoint is the ORR (objective response rate), based on local investigator assessment, per RECIST 1.1. | 6 months after study treatment initiation
  the ORR (objective response rate), defined as the proportion of patients who have achieved a complete response (CR) or partial response (PR) within the first 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Paule SABLIN, MD, PhD, Principal Investigator — Institut Curie
Locations (4):
- France (4):
  - CLCC F.Baclesse Caen, Caen
  - Institut Curie, Paris
  - Institut de Cancerologie de l'Ouest- ICO, Saint-Herblain
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Background] 1.Ezzalfani M. et al. The role of the expansion cohort in phase I trials in oncology: guidelines of the phase I HUB. Bull Cancer. 2015 Jan;102(1):73-82. doi:10.1016/j.bulcan. 2014.10.001. Epub 2015 Jan 2. Review. French. 2.M3(R2) guideline : Nonclinical Safety Studies for the Conduct of Human Clinical Trials and Marketing Authorization for Pharmaceuticals 3.ICH S9 - Nonclinical Evaluation for Anticancer Pharmaceuticals EMEA/CHMP/ICH/646107/2008 4.Masini et al. Histamin-releasing properties of polysorbate 80 in vitro and in vivo: correlation 1254 with its hypotensive action in the dog. Agents Actions 1985 Sep; 16(6):470-7. 5.Guideline on repeated dose toxicity - CPMP/SWP/1042/99 Rev 1 6.Storer B.E. Design and Analysis of Phase I Clinical Trials. Biometrics, Vol. 45, No. 3 (Sep., 1989), pp. 925-937. 7.Seshan V.E. et al. Clinical Trial Design and Data Analysis Functions, Package clinfun, version 1.0.15 (Apr 2018)